CLINICAL TRIAL: NCT02321787
Title: Utility of Ultrasonography for Confirmation of Successful Caudal Epidural Injection
Brief Title: Ultrasonography for Confirmation of Caudal Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #2015-16004
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Pain, Postoperative
Keywords: Anesthesia, Caudal; Ultrasonography
MeSH Terms: conditions — Pain, Postoperative | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Methods of Assessment (No Intervention): The caudal block will be done using traditional means of assessment, not confirmed by ultrasound.
- Ultrasound for Confirmation (Experimental): The caudal block will be performed utilizing ultrasound as an additional method of assessment for successful block (in addition to all traditional means of assessment).
  Interventions: Procedure: Ultrasound for confirmation of successful caudal block

INTERVENTIONS:
Procedure: Ultrasound for confirmation of successful caudal block — Use of ultrasound for confirmation of successful caudal block
  Arms: Ultrasound for Confirmation

SUMMARY:
The purpose of our study is to evaluate whether utilizing ultrasound assessment during caudal epidural injection can reliably identify unrecognized and unsuccessful nerve blocks during the procedure, guide proper technique, and alter pain management outcome measurements for patients.

Patients will be randomized to a group either undergoing caudal injection by a trainee using typical techniques or by using typical techniques in addition to ultrasound for confirmation of successful injection. The patients enrolled in this study will have the same intraoperative care, in line with the standard of care. Data will be collected intraoperatively and postoperatively on pain scores, time for performance of caudal block, and perceived success of the block. There will be no direct benefit to the patients enrolled in this study, but future patients may benefit from the use of ultrasound for the confirmation of a successful block.

DETAILED DESCRIPTION:
Caudal epidural injection is the most commonly performed regional anesthetic procedure in infants and children and is used to provide perioperative analgesia for many lower abdominal, lower extremity, and urological procedures. Utilizing sterile technique, a needle is advanced through the sacral hiatus and local anesthetic is injected into the epidural space. Local anesthetic spreads cranially and results in significant sensory (+/- motor) blockade, depending on local anesthetic concentration and volume1. Recent studies have used ultrasound to assess cranial spread during caudal blockade, specifically evaluating how speed of injection and different volumes can affect cranial spread2,4. Other studies have investigated redistribution and secondary spread after initial injection of local anesthetic by utilizing ultrasound assessment of the epidural space3.

Although no current standard exists for confirming successful caudal epidural injection, several findings may indicate a proper needle position and can predict successful block5. Some of these findings include: tactile appreciation of the "pop" through the sacrococcygeal ligament, negative blood or cerebrospinal fluid aspiration, negative test dose, appropriate resistance during injection, no subcutaneous swelling during injection, no motor or hemodynamic response to skin incision, and no need for administration of supplemental analgesics. Although several studies have shown that real-time ultrasound guidance can be used during needle insertion for caudal block, this does not guarantee adequate cranial spread and may be technically challenging for a trainee performing the block. Furthermore, many of the tactile findings that indicate successful entry into the appropriate space can only be appreciated by the trainee, not the supervising anesthesiologist, which complicates supervision of this technique. At present, difficulty in reliably predicting block failure may lead to overuse of narcotics to prevent pain in patients with potentially failed blocks or could lead to inadequate analgesia in patients too young to reliably communicate their pain level.

The purpose of our study is to evaluate whether utilizing ultrasound assessment during caudal epidural injection can reliably identify unrecognized and unsuccessful nerve blocks during the procedure, guide proper technique, and alter pain management outcome measurements for patients.

The proposed study will not change the current practice with regard to patient selection for caudal epidural injection and will not change the performance of the procedure itself. This study may impact the practice of general pediatric anesthesiologists by providing evidence that ultrasound is a useful tool for determining successful caudal epidural injection, may help identify unrecognized failed blocks earlier and will evaluate which level(s) of anesthesia training would most benefit from this assessment tool.

Patients will be randomized using pre-made folders containing an assignment to either the control group or study group. In the study group, ultrasound will be utilized in the caudal block to confirm placement. In the control group, the caudal block will be done without ultrasound to assist with caudal epidural injection. In the operating room, once the anesthesia team is prepared to begin the caudal epidural injection, the patient will be placed in the lateral decubitus or prone position, with knees and hips flexed. The attending for the caudal block will mark the site on the patient per the site marking policy at Lurie Children's; this is not necessarily the attending of record for the remainder of the case. Once the sacrum is prepped, the anesthesia provider will proceed with the caudal epidural injection in the usual fashion. The injected solution will be 1 mL/kg of 0.2% ropivacaine with 1:200k epinephrine, rounded up to the next mL, which is consistent with the current standard practice at Lurie Children's. After injection of test dose (10% of the total block volume), a one-minute pause will begin to assess for a response. During this pause, prior to injection of the remaining dose of local anesthetic, a 13-6 MHz, linear ultrasound probe with a sterile covering and ultrasound gel will be placed over the patient's lumbar spine, cranial to the point of entry for the caudal block. The caudal block needle insertion site and sterile field will be observed and undisturbed. The ultrasound probe will be positioned paramedian along the non-dependent side of the spine, obtaining a long axis view of the epidural and intrathecal space. The cephalad end of probe will be placed at the level of the iliac crest. Once the ultrasound probe is positioned properly and the one-minute pause has finished, the remaining dose of local anesthetic will be administered by the anesthesia provider as an ultrasound clip of epidural spread is visualized.

The supervising attending anesthesiologist will be one of those listed in the personnel form. In either group, the attending anesthesiologist will coach the resident to help guide them to success based on the standards of care with this block. In the control group, if it is felt that the trainee is unable to safely and successfully perform the block based on typically utilized methods of assessment (injection pressure, needle appearance, subcutaneous swelling) then the attending will take over the block, consistent with current practice at Lurie Children's. In the study group, the attending will continue to use traditional methods of assessment but will also utilize the ultrasound to assess block success and may either take over the block at the time injection has been determined to be unsuccessful or may redirect the trainee to success in their performance of the block.

As part of the research protocol, the primary anesthesia team should avoid giving the patient other analgesic medications prior to the time of incision. Additionally, the anesthesia team should have the patient at 1 MAC of sevoflurane and avoid using nitrous oxide, at the time of incision. After incision, all anesthetic decisions will be at the discretion of the attending anesthesiologist of record in the operating room.

Data will be collected on the level of training of the physician performing the procedure, the proceduralist's experience level, findings during the procedure, and their confidence level of block success. Subsequent data will be collected on response to skin incision and need for supplemental analgesia. In the recovery room, a pain score will be assessed at the time of phase 1 recovery discharge. Recovery room staff will be advised to only give analgesic medications, standardized to 0.05 mg/kg of morphine, if pain is rated at > 4 on the rFLACC scale, appropriate to the patients' age. The ultrasound probe placement, image acquisition, survey administration, pre-incision anesthetic standardization, and recovery room analgesic administration threshold are the only research-related procedures. All elements of patient care described above, including withholding additional analgesics before incision, are consistent with the current standard of care and standard practices at Lurie Children's. The length of the study visit will be from the time of operation until PACU discharge, with the intervention only taking place during the operation.

Caudal analgesia will be rated successful if 2 conditions are fulfilled: (1) the procedure was performed without any physical assistance by the supervisor, with verbal comments and suggestions allowed, and no more than 3 passes with the needle through the skin needed, and (2) clinical success of the block. Clinical failure will be defined as need for opioid supplementation or increased concentration of volatile anesthetic in response to clinical signs of insufficient analgesia including increases in heart rate, blood pressure, movement of patient, or other signs of stress at incision or during the procedure. The attending anesthesiologist will predict whether the caudal block was successful based on clinical indicators alone in the control group and based on ultrasound findings in the study group. This assessment of confidence in the block must be made before emergence from anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Under the age of eight
* 20kg or less
* Who are undergoing lower abdominal, lower extremity orthopedic, or urological procedures in the operating room at Ann & Robert H. Lurie Children's Hospital of Chicago (Lurie Children's) and will have a caudal epidural injection performed by an anesthesia resident physician prior to surgical incision
* Children will be the sole patient population for this study

Exclusion Criteria:

* Patients will be excluded if their ultrasound images are deemed inadequate for evaluation of epidural injection
* The caudal injection is abandoned after unsuccessful attempts
* The surgical incision is at or above the umbilicus

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Rate of block success in traditional group versus intervention (ultrasound) group | 4 hours
  Success in the ultrasonographic group will be estimated by ultrasound spread and in the traditional group by heart rate, need for additional medications, and pain scores.

SECONDARY OUTCOMES:
Opioid Administration | 4 hours
  Opioid administration will be compared between the control and intervention groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Lundblad M, Lonnqvist PA, Eksborg S, Marhofer P. Segmental distribution of high-volume caudal anesthesia in neonates, infants, and toddlers as assessed by ultrasonography. Paediatr Anaesth. 2011 Feb;21(2):121-7. doi: 10.1111/j.1460-9592.2010.03485.x. Epub 2010 Dec 15. PMID 21159024
- [Background] Triffterer L, Machata AM, Latzke D, Willschke H, Rebhandl W, Kimberger O, Marhofer P. Ultrasound assessment of cranial spread during caudal blockade in children: effect of the speed of injection of local anaesthetics. Br J Anaesth. 2012 Apr;108(4):670-4. doi: 10.1093/bja/aer502. Epub 2012 Feb 6. PMID 22315328
- [Background] Lundblad M, Eksborg S, Lonnqvist PA. Secondary spread of caudal block as assessed by ultrasonography. Br J Anaesth. 2012 Apr;108(4):675-81. doi: 10.1093/bja/aer513. Epub 2012 Feb 6. PMID 22315327
- [Background] Brenner L, Marhofer P, Kettner SC, Willschke H, Machata AM, Al-Zoraigi U, Lundblad M, Lonnqvist PA. Ultrasound assessment of cranial spread during caudal blockade in children: the effect of different volumes of local anaesthetics. Br J Anaesth. 2011 Aug;107(2):229-35. doi: 10.1093/bja/aer128. Epub 2011 Jun 3. PMID 21642642
- [Background] Raghunathan K, Schwartz D, Connelly NR. Determining the accuracy of caudal needle placement in children: a comparison of the swoosh test and ultrasonography. Paediatr Anaesth. 2008 Jul;18(7):606-12. doi: 10.1111/j.1460-9592.2008.02529.x. PMID 18616491
- [Background] Riccabona M. Basics, principles, techniques and modern methods in paediatric ultrasonography. Eur J Radiol. 2014 Sep;83(9):1487-94. doi: 10.1016/j.ejrad.2014.04.032. Epub 2014 May 10. PMID 24932845
- [Background] Schuepfer G, Konrad C, Schmeck J, Poortmans G, Staffelbach B, Johr M. Generating a learning curve for pediatric caudal epidural blocks: an empirical evaluation of technical skills in novice and experienced anesthetists. Reg Anesth Pain Med. 2000 Jul-Aug;25(4):385-8. doi: 10.1053/rapm.2000.7590. PMID 10925935